CLINICAL TRIAL: NCT05957289
Title: Effect of Metaverse-based Multidimensional Rehabilitation Intervention on Quality of Life and Fear of Recurrence in Colorectal Cancer Survivors - a Pilot Study
Brief Title: Multidimensional Rehabilitation Intervention in Colorectal Cancer Survivors - a Pilot Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qu Shen (Other)
Collaborators: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor-Investigator, Qu Shen, Associate Professor, Xiamen University
Organization: Xiamen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: XiamenUSQ
Record Dates: First submitted 2023-07-13; First posted 2023-07-24 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Rehabilitation; Colorectal Cancer Survivor; Quality of Life; Pilot Study
Keywords: Colorectal cancer survivor; Rehabilitation; Quality of Life; Fear of cancer recurrence; Lifestyle; Home-based

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multidimensional rehabilitation group (Experimental): The intervention is based on the behavior change wheel and includes dietary intervention, exercise intervention, psychological support, and behavior management. Through various methods such as training, education, and motivation, the patient's ability, opportunities, and motivation will be increased, thereby promoting healthy behavior.
  Interventions: Behavioral: multidimensional rehabilitation

INTERVENTIONS:
Behavioral: multidimensional rehabilitation — Multidimensional lifestyle interventions

SUMMARY:
A metaverse-based multidimensional rehabilitation program will be implemented for colorectal cancer survivors who have undergone curative surgery and adjuvant therapy. The intervention is based on the behavior change wheel and includes dietary intervention, exercise intervention, psychological support, and behavior management. Through various methods such as training, education, and motivation, the program aims to enhance the patients' functional ability, opportunities, and motivation, thereby promoting healthy behavior. Outcome measures include quality of life, fear of recurrence, and adoption of a healthy lifestyle. The intervention period is 4 weeks, with evaluations conducted at baseline and week 4 of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing adjuvant therapy after curative surgery for colorectal cancer.;
* Age 18 years old and under 65 years old, estimated survival period ≥ 6 months;
* PG-SGA (Patient-Generated Subjective Global Assessment) score less than 4.
* be able to walk without assistance;
* Conscious and intellectually normal;
* Voluntarily participate in the research of this topic and provide the consent form for medical record review;
* Mobile phones can be used.

Exclusion Criteria:

* Patients with multiple cancers.
* Tumors not completely resected.
* Patients with severe psychological disorders, severe visual or hearing impairments, or other conditions that hinder intervention.
* Patients with severe complications such as short bowel syndrome, Crohn's disease, ulcerative colitis, diverticulitis, previous stroke, congestive heart failure or edema, liver or kidney failure, or other conditions that affect patient compliance.
* In addition to colorectal cancer or any other diseases deemed unsuitable for participation by the researchers, patients with severe heart, liver, lung, or kidney diseases.
* Patients with special dietary requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events | 4th week
  Record the occurrence of adverse events, including nausea, vomiting, pain, etc.
Adherence | 4th week
  The number of days per week that participants complied with the protocol will be recorded over a 4-week period.
Viability | 4th week
  Record the number and reasons for loss to follow-up
Chinese version of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) | Change from Baseline at 4 weeks
  This Scale was developed to measure the quality of life of patients with cancer. It includes 30 questions and three sub-dimensions: General Well-Being, Functional Difficulties, and Symptom Control. The maximum score on the scale is 100, and the minimum is 0. High scores on the functional sub-dimension indicate good/healthy functional status, high scores on the symptom sub-dimension indicate high levels of symptoms and/or problems, and high scores on the global health status/quality of life sub-dimension indicate good quality of life.
Fear of Progression Questionaire-Short Form (FoP-Q-SF) | Change from Baseline at 4 weeks
  The FoP-Q-SF was developed by German scholar Herschbach in 2005 in people such as diabetes, rheumatic diseases and cancer, to measure patients' fear of disease progression or recurrence, a total of 7 dimensions, 43 entries, Cronbach's α is 0.7. It is a single-dimensional scale with a total of 12 items, using the Liket 5-level scoring method, the score range is 12~60, the higher the score, the higher the level of fear.

SECONDARY OUTCOMES:
Lifestyle | Change from Baseline at 4 weeks
  Assessments of lifestyle behaviors will be conducted using a self-developed behavior scale, focusing on the frequency of behaviors such as diet and smoking.
The International Physical Activity Questionnaire (IPAQ) | Change from Baseline at 4 weeks
  The International Physical Activity Questionnaire (IPAQ) is a commonly used tool for assessing individuals' levels of physical activity in their daily lives. It aims to measure individuals' physical activity over the past 7 days, including overall physical activity levels and the frequency of activities.
30-second Chair Sit-To-Stand (30-s STS) | Change from Baseline at 4 weeks
  Ability to test mobility and posture transposition. Using a chair without armrests, the number of times the participant could change from a sitting state (leaning back on the chair with both feet on the ground) to fully standing within 30 s was counted. Two tests were performed, with 1 min of rest in between, and the average value was rounded to the nearest value.
BMI | Change from Baseline at 4 weeks
  BMI reflects the patient's nutritional status and physical fitness.
Semi-structured interviews | 4th week
  After the intervention, semi-structured interviews were conducted with the participants. The main topics covered included the benefits and adverse reactions of the multidimensional rehabilitation intervention, factors that facilitated or hindered participation in the multidimensional rehabilitation, and the pros and cons of the metaverse platform.

IPD SHARING:
Plan to Share IPD: Yes